CLINICAL TRIAL: NCT04784598
Title: Effects of Insoles Adapted in Flip-flop Sandals in People With Heel Pain: a Randomized, Double-blind Clinical, Controlled Study
Brief Title: Insoles Adapted in Flip-flop Sandals in People With Heel Pain
Acronym: Heelpain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, PT, PhD., Adjunct Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFRNheelpain
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Heel Pain Syndrome; Heel

STUDY DESIGN:
Intervention Model Description: Group 1- (n=40) The participant allocated to the insoles group adapted to flip-flops and classified as having a neutral foot according to the FPI-6 will receive a flip-flop with a horseshoe-type foot element on both feet to maintain symmetry between the limbs.
  If the participant is classified with the foot pronated or supinated, only the painful foot will be modified since the symmetry of the limbs will not be modified. Participants with pronated foot will receive the medial wedge as a pedal element; already the participants with supinated foot, the lateral wedge. All elements will be 3mm and produced with EVA Shore 32.
  • Group 2- The control group (n=40) will receive a slipper with a 2.5mm EVA cover (Shore A 32) identical to the one used by the intervention group, but without corrective par.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group 1- The intervention group I will receive a customized strip slipper with a 3mm EVA horseshoe piece (Shore A 32). And 2.5mm EVA cover (Shore A 28).
  Interventions: Other: Insoles adapted in flip-flop sandals
- Sham group (Sham Comparator): Group 2- The control group will receive a slipper with a 2.5mm EVA cover (Shore A 32) identical to the one used by the intervention group, but without corrective par
  Interventions: Other: Insoles adapted in flip-flop sandals

INTERVENTIONS:
Other: Insoles adapted in flip-flop sandals — participants of both groups individually received a pair of customized flip-flop sandals, with or without foot pieces, covered with smooth synthetic leather

SUMMARY:
Introduction: Persistent hindfoot pains are very common and prevalent complaints in the Brazilian population. One of the treatments recommended for these conditions in the literature is the use of insoles. However, to use this resource it is necessary that the individual wear closed shoes and this is an obstacle to treatment in cities with hot climate. Thinking about an alternative treatment, the customized slippers with the corrective elements of the insoles can be an alternative to increase adherence to this type of treatment. Objective: To compare different types of hindfoot elements in insoles adapted in slippers in individuals with persistent hindfoot pain.

DETAILED DESCRIPTION:
Methodology: This is a protocol for a controlled, randomized, blinded clinical trial. Eighty participants with persistent hindfoot pain will be evaluated and randomized into two intervention groups: insoles adapted to flip-flops and flip-flops with sham insole. The evaluations will be carried out at baseline (T0), after six (T6) and twelve weeks (T12) of the use of flip-flops, in addition to the follow-up that will be carried out four weeks after the end of the intervention (T16). The primary outcome will be pain, using the Numerical Pain Scale and the secondary outcomes will be: foot function, using the Foot Function Index questionnaire, functional capacity in walking, using the Six-Minute Walk Test and pain catastrophizing using the Scale. of Pain Catastrophizing. Statistical analysis: Data will be analyzed by T-student, Mann-Whitney and repeated measures ANOVA tests and will be analyzed by intention to treat. Ethics and disclosure: This protocol was approved by the Ethics Committee of UFRN/FACISA (number 4,018,821). The results of the study will be disseminated to participants and submitted to a peer-reviewed journal and scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes, aged 18 to 65 years;
* Persistent heel pain for at least three months based on self-reported criteria: heel pain accompanying the first steps in the morning, after a period of inactivity, and/or during prolonged weight-bearing;
* Pain intensity between 3 and 8 points, according to the Numerical Rating Scale (NRS) [22];
* Individuals who can wear flip-flop sandals for at least four hours per day for 12 weeks.

Exclusion Criteria:

* Clinical diagnosis of neuropathic pain or neurodegenerative disorders, persistent heel pain due to rheumatic conditions, and previous ankle and foot surgeries;
* Physical therapy treatment in the last three months;
* Corticosteroid injection into feet in the last six months;
* inability to answer study-related questionnaires;
* Individuals scheduled to travel in the next six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Numerical pain intensity scale - NPS | baseline, 6 weeks after, 12 weeks after, 16 weeks folow up
  Pain intensity will be evaluated with the 10-point Numerical Pain Rating Scale, where 0 is "pain-free" and 10 is "maximum pain.

SECONDARY OUTCOMES:
Change in Foot function - FFI | baseline, 6 weeks after, 12 weeks after, 16 weeks folow up
  Brazilian version of the Foot Function Index questionnaire.15 This questionnaire aims to evaluate the functionality of the foot and is divided into three subscales, which are pain, difficulty and functional limitation. The outcome of all domains was summed and divided by three to achieve the final result of the questionnairewhich can vary from 0% to 100%, and are proportional to functional impairment of the limb.The higher the percentage, the greater the functional alteration presented by the patient
Change in Functional capacity - 6MWT | baseline and 12 weeks after
  For this test, the participant walked at full speed for 6minutes along a 30-m lane, and the total distance was recorded.
Change in Pain Catastrophizing Scale (PCS) | baseline and 12 weeks after
  Self-administered questionnaire composed of 13 items in which the individual reports the degree of thought or feeling on a 5-point Likert scale. The instrument has three subscales (hopelessness, magnification, and rumination), and the total score (0 to 52 points) is obtained by summing items. The higher the value, the greater the level of catastrophizing
Expectation for treatment | baseline
  The scale assesses the expectations of individuals at the beginning of the study regarding treatment received. The question "Do you think that with flip-flop sandals you will" (1) get very worse, (2) get a little worse, (3) neither improve nor get worse, (4) improve a little, or (5) improve a lot. This scale will be applied only in the first (T0) assessment
Satisfaction with treatment | 16 weeks after
  The scale will assess perceptions of the individual on the effects of treatment through the following question: "After using flip-flop sandals with insoles are you feeling" (1) much worse, (2) a little worse, (3) neither better nor worse, (4) a little better, or (5) much better

CONTACTS AND LOCATIONS:
Locations (1):
- Marcelo Cardoso de Souza, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Result] Costa ARA, de Almeida Silva HJ, Mendes AAMT, Scattone Silva R, de Almeida Lins CA, de Souza MC. Effects of insoles adapted in flip-flop sandals in people with plantar fasciopathy: a randomized, double-blind clinical, controlled study. Clin Rehabil. 2020 Mar;34(3):334-344. doi: 10.1177/0269215519893104. Epub 2019 Dec 6. PMID 31808352
- [Derived] Fagundes MG, Mendes AAMT, Bezerra VF, Freitas WRMS, Scattone Silva R, Pontes-Silva A, Barbosa GM, Cardoso de Souza M. Effects of insoles adapted in flip-flop sandals in patients with persistent plantar heel pain: A sham-controlled randomised trial. Clin Rehabil. 2024 Nov;38(11):1466-1480. doi: 10.1177/02692155241267991. Epub 2024 Aug 2. PMID 39094377
- [Derived] Fagundes MG, Teixeira Mendes AAM, Barbosa GM, de Souza MC. Effects of insoles adapted in flip-flop sandals for persistent heel pain: a protocol for a sham-controlled randomised trial. BMJ Open. 2022 Nov 7;12(11):e062523. doi: 10.1136/bmjopen-2022-062523. PMID 36343988